CLINICAL TRIAL: NCT06362421
Title: Proof of Concept Assay Development of Point of Care Saliva Testing for High Risk-HPV Oral Cavity and Pharynx Cancers
Brief Title: Saliva Testing for High-Risk Human Papillomavirus Infection Oral Cavity and Pharynx Cancer
Status: Withdrawn | Type: Observational
Why Stopped: PI not moving forward with study at our institution
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: InnoTech Precision Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00115786; ONC-HN-2402 (Other: WFBCCC)
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma; Human Papillomavirus Infection
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Papillomavirus Infections | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment naive patients with HPV+ OPSCC: Participants will receive a pre-study visit and pre-radiation dental evaluation.
  Interventions: Genetic: Pre-Radiation Dental Evaluation/Sample Collection; Other: Pre-Study Visit
- Control Group - Healthy subjects without cancer: Participants will receive a pre-study visit and oral medicine consultation visit.
  Interventions: Other: Pre-Study Visit; Genetic: Oral Medicine Consultation Visit/Sample Collection

INTERVENTIONS:
Genetic: Pre-Radiation Dental Evaluation/Sample Collection — Collection of saliva samples and mouth swabs and pre-cancer dental evaluation by study staff. Unstimulated saliva will be collected then a buccal swab sample will be obtained. Participants will be asked to rinse their mouth with water, wait 10 minutes, then 1-2 mL of unstimulated saliva will be captured into sterile centrifuge tube. Next, a buccal swab sample will be collected using a sterile cotton swab and immediately placed in a transport tube containing buffer (Tris with low EDTA)
  Groups: Treatment naive patients with HPV+ OPSCC
Other: Pre-Study Visit — Collection of vital signs, medical history and current medications
Genetic: Oral Medicine Consultation Visit/Sample Collection — Collection of saliva samples and mouth swab, complete oral medicine consultation by study staff. Unstimulated saliva will be collected then a buccal swab sample will be obtained. Participants will be asked to rinse their mouth with water, wait 10 minutes, then 1-2 mL of unstimulated saliva will be captured into sterile centrifuge tube. Next, a buccal swab sample will be collected using a sterile cotton swab and immediately placed in a transport tube containing buffer (Tris with low EDTA)
  Groups: Control Group - Healthy subjects without cancer

SUMMARY:
The purpose of this research study is to determine if saliva and oral swab samples can be used to detect human papillomavirus in patients with cancer. In this study, the methods required to detect human papillomavirus will be developed and tested in samples collected from patients with oropharyngeal squamous cell carcinoma and compared to samples collected from participants without cancer.

DETAILED DESCRIPTION:
To validate the detection of human papillomavirus 16 and 18 and reference gene ACTB in saliva and buccal swab samples obtained from patients with oropharyngeal squamous cell carcinoma (OPSCC) using the LAMP/CRISPR/electrochemical workflow.

ELIGIBILITY:
Inclusion Criteria (Patients with Cancer);

* Patients must have histologically confirmed oropharyngeal squamous cell carcinoma without prior treatment. A pathology report should be referenced/available.
* Patients with p16 positive oropharyngeal squamous cell carcinoma.
* Age 39 to 59 years.
* Ability to understand and the willingness to sign an IRB-approved informed consent document directly.

Inclusion Criteria (Healthy Subjects)

* Age 39 to 59 years.
* Ability to understand and the willingness to sign an IRB-approved informed consent document directly.

Exclusion Criteria (Patients with Cancer)

* Patients with diagnoses of other cancers.
* Patients with current or previous diagnosis with HPV+ infection status for cervical cancer or other cancers.

Exclusion Criteria (Healthy Subjects)

* Previous diagnosis of cervical cancer or other cancers.
* Presence of known active oral infections of viral, fungal, or bacterial etiology except for gingivitis, periodontitis, or periapical abscess. Participants with known gingivitis, periodontitis, or periapical abscess are included.

Ages: 39 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Head and Neck oncology team and navigators, as well as tumor board meetings, will be leveraged to identify and recruit newly diagnosed patients.
  Participants in the healthy control group will be identified and recruited and enrolled after patients in the research cohort (those with OPSCC) participants have been enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Sensitivity for Detection of HPV 16, 18 and gene ACTB | Up to 2 years
  The sensitivity of the LAMP/CRISPR/electrochemical workflow for detection of HPV 16, 18, and reference gene ACTB will be measured using patient samples with a 95% Clopper Pearson Exact Binomial confidence interval for the estimated sensitivity (or specificity) will have a lower bound of 83% if the observed sensitivity (or specificity) is 95%. For each of these estimates investigators will examine the proportion and the corresponding 95% Clopper Pearson exact binomial confidence interval.
Number of Participants with Specificity Detection of HPV 16, 18 and gene ACTB | Up to 2 years
  The specificity of the LAMP/CRISPR/electrochemical workflow for detection of HPV 16, 18, and reference gene ACTB will be measured using patient samples with a 95% Clopper Pearson Exact Binomial confidence interval for the estimated sensitivity (or specificity) will have a lower bound of 83% if the observed sensitivity (or specificity) is 95%. For each of these estimates investigators will examine the proportion and the corresponding 95% Clopper Pearson exact binomial confidence interval.
Overall Accuracy - All Participants | Up to 2 years
  For estimating overall accuracy (using all patients with n=80), the confidence interval will have a lower bound of 88% if the accuracy is at least 95%. For each of these estimates investigators will examine the proportion and the corresponding 95% Clopper Pearson exact binomial confidence interval.

IPD SHARING:
Plan to Share IPD: No